CLINICAL TRIAL: NCT06634693
Title: Accuracy of Pulse Oximeters with Profound Hypoxia
Brief Title: Controlled Desaturation Study for TipTraQ SpO2 Performance Validation
Status: Completed | Type: Observational
Sponsor: PranaQ Pte. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: TipTraQ SpO2 validation study; 21-35637 (Registry Identifier: Accuracy of pulse oximeters with profound hypoxia)
Record Dates: First submitted 2024-10-03; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Hypoxia
Keywords: SpO2
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Heathy adult: healthy adult without pulmonary or cardiovascular disease

SUMMARY:
The objective is to validate the performance of SpO2 measurement of the TipTraQ by comparing it with measurement from an artery blood sample of a healthy volunteer in a controlled desaturation study. The overall framework of the validation process followed Annex EE.2 of ISO 80601-2-61:2019.

DETAILED DESCRIPTION:
The TipTraQ, is a finger-based wearable for aiding OSA diagnosis at home that consists of a sensor placed on a fingertip. PPG data are produced by a reflective emitter and photodetector elements from one of the fingertips. TipTraQ Companion app can read and record the PPG signals from the TipTraQ Sensor and further transmit the data to TipTraQ Cloud.

The overall framework is a controlled desaturation study follows the Annex EE.2 of ISO 80601-2-61:2019. A radial arterial cannula was placed in each subject's left or right wrist for blood sampling and monitoring blood pressure. Each subject had two control blood samples taken at the beginning of each experiment while breathing room air. Hands with pulse oximeters were maintained motionless on arm boards. Hypoxia was then induced to different and stable levels of oxyhemoglobin saturation (between 70-100%) by having subjects breathe mixtures of nitrogen, air, and carbon dioxide controlled by the study physician by adjusting gas flows with valves according to breath-by-breath estimates of oxygen saturation calculated from end-tidal PO2 and PCO2. Each plateau level of oxyhemoglobin saturation was maintained for at least 30 seconds or until reference pulse oximeter readings were stable. During the procedure, the subject is under stationary status. Two arterial blood samples were then obtained approximately 30 seconds apart. Each stable plateau, therefore, was maintained for at least 60 seconds with SpO2 fluctuating by less than 2-3%. The plateaus were nominally at 100%, room air saturation, 93%, 90%, 87%, 85%, 82%, 80%, 77%, 75% and 70%. At least 200 data points were collected for each type of oximeter and probe combination studied.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have the ability to understand and provide written informed consent
* A participant is an adult 18-50 years of age
* Participant must be willing and able to comply with study procedures and duration
* Participant is a non-smoker or who has not smoked within 2 days before the study.

Exclusion Criteria:

* Participant is considered as being morbidly obese (defined as BMI >39.5)
* Compromised circulation, injury, or physical malformation of fingers, toes, hands, ears, forehead/skull, or other sensor sites would limit the ability to test sites needed for the study. Tattoos in the optical path would limit the ability to test sites needed for the study.
* Participants with known respiratory conditions
* Uncontrolled/severe asthma
* pneumonia/bronchitis
* shortness of breath / respiratory distress, unresolved respiratory or lung surgery, emphysema, COPD, lung disease
* Recent COVID (last 2 months)
* Participants with self-reported heart or cardiovascular conditions
* chest pain (angina)
* heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia
* previous heart attack
* blocked artery
* congestive heart failure (CHF)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults without respiratory or heart diseases
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
SaO2 | During the controlled desaturation study, within 1 day
  oxygen saturation of arterial blood sample measured by blood gas analysis
SpO2 | During the controlled desaturation study, within 1 day
  Peripheral blood oxygen saturation measured through plethysmography(PPG)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Bickler, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Medical Center at Parnassus, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No